CLINICAL TRIAL: NCT06413342
Title: Sintilimab After Concurrent Chemoradiotherapy in Elderly Patients With Unresectable Esophageal Squamous Cell Carcinoma: A Randomized, Multi-center Phase II Clinical Trial
Brief Title: Sintilimab After Concurrent Chemoradiotherapy in Elderly Patients With Esophageal Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yang Yang, Clinical Professor, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2023-1237
Record Dates: First submitted 2024-05-08; First posted 2024-05-14 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Esophageal Cancer; Chemoradiotherapy; Sintilimab; Immunotherapy; Elderly Patients
MeSH Terms: conditions — Esophageal Neoplasms | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sintilimab group (Experimental): Patients in treatment group receive sintilimab (for patients with a weight <60 kg: 3 mg/kg IV on Day 1 every 3 weeks; for patients with a weight ≥60 kg: 200 mg IV on Day 1 every 3 weeks) .
  Interventions: Drug: Sintilimab
- Observation group (No Intervention): Patients in the observation group receive regular follow-up and observation.

INTERVENTIONS:
Drug: Sintilimab — Patients should receive their first dose of sintilimab within 42 days after completing the final radiotherapy session and continue treatment until disease progression, occurrence of intolerable toxicity, loss to follow-up, death, or as determined by the investigator, whichever comes first. The maximum duration of sintilimab treatment is 12 months (from the initiation of therapy). No other anti-tumor therapies are permitted during the treatment period.
  Arms: Sintilimab group

SUMMARY:
This trial is a prospective, randomized, controlled, multicenter, phase II clinical study to evaluate the efficacy and safety of sintilimab as consolidation therapy in elderly patients with esophageal cancer who did not progress after concurrent chemoradiotherapy.

Patients aged 70-85 years with esophageal squamous cell carcinoma who did not progress after concurrent chemoradiotherapy and meet the inclusion criteria will be stratified according to MRD status (positive vs negative) and randomized in a 1:1 ratio into two groups: the treatment group receiving sintilimab (for patients with a weight <60 kg: 3 mg/kg IV on Day 1 every 3 weeks; for patients with a weight ≥60 kg: 200 mg IV on Day 1 every 3 weeks) and the observation group receiving regular follow-up. Patients should receive the first dose within 42 days after completing the last radiotherapy session and continue treatment until disease progression, intolerable toxicity, loss to follow-up, death, or other circumstances where the investigator determines treatment should be discontinued, whichever occurs first. The maximum duration of sintilimab treatment is 12 months (from the start of treatment), while the observation group will be followed up every 3 months for at least one year. No other anti-tumor treatments are allowed during the study period. The study aims to compare the effects of the two treatment modalities on progression-free survival, overall survival, tumor response, toxicity reactions, and quality of life in elderly patients with esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed squamous cell carcinoma of the esophagus, clinically staged before treatment (8th edition of the UICC/AJCC TNM staging system for esophageal squamous cell carcinoma) as stage II-IVb (cT1N2-3M0-1, cT2-4bN0-3M0-1, M1 limited to supraclavicular lymph node metastasis).
2. Candidates for curative esophageal cancer surgery who are unable to tolerate surgery or refuse surgery.
3. Age 70 to 85 years.
4. ECOG performance status of 0-1.
5. The minimum technical standard for radiotherapy is intensity-modulated radiotherapy (IMRT). The total dose of radiotherapy is 54Gy ± 10%.

   Note: It is recommended that study centers conduct screening within 14 days after subjects complete synchronous chemoradiotherapy.
6. Concurrent chemotherapy regimen: Single-agent S-1 70mg/m2, days 1-14 and 29-42, synchronized with radiotherapy for 14 days or longer.
7. The last cycle of chemotherapy must end before or concurrently with the last session of radiotherapy. Consolidation chemotherapy after radiotherapy is not allowed, and chemotherapy before chemoradiotherapy is not accepted. Patients who have not progressed after chemoradiotherapy, including complete response (CR), partial response (PR), and stable disease (SD), can be enrolled in this study.
8. Except for hearing loss, hair loss, and fatigue, all toxicities from previous anti-tumor treatments must have recovered to grade ≤1 (according to the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] v5.0) or baseline level before enrollment.
9. The first dose of study medication must be administered within 42 days after completion of chemoradiotherapy.
10. No esophageal perforation or active esophageal bleeding, no significant invasion of the trachea or major blood vessels in the chest. No interstitial pneumonia or history of interstitial pneumonia. FEV1 ≥ 0.8L.
11. Expected survival ≥ 3 months.
12. Laboratory criteria:

    1. Serum hemoglobin ≥ 90g/L, platelets ≥ 100 × 10^9/L, absolute neutrophil count ≥ 1.5 × 10^9/L.
    2. Serum creatinine ≤ 1.5 times the upper limit of normal (ULN) or creatinine clearance ≥ 40 mL/min.
    3. Serum bilirubin ≤ 1.5 times ULN, AST (SGOT) and ALT (SGPT) ≤ 2.5 times ULN, alkaline phosphatase ≤ 5 times ULN.
    4. International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN (patients on stable doses of anticoagulant therapy such as low molecular weight heparin or warfarin with an INR within the expected therapeutic range for anticoagulant therapy can be screened).
13. Patients must sign formal informed consent forms indicating their understanding that this study complies with hospital policies and ethical requirements.

Exclusion Criteria:

* 1. Patients who underwent surgical resection for esophageal cancer prior to the start of this trial or have previously received treatment with immune checkpoint inhibitors such as anti-PD-1/PD-L1 or CTLA-4 inhibitors.

  2. Patients staged as cT1-3N1-2M0, deemed suitable for surgical resection, and requiring surgery.

  3. Experience disease progression after chemoradiotherapy. 4. High risk of gastrointestinal bleeding, esophageal fistula, or esophageal perforation.

  5. History of interstitial lung disease, non-infectious pneumonia, pulmonary fibrosis, or other uncontrolled acute pulmonary conditions.

  6. Poor nutritional status, with a BMI less than 18.5kg/m2, or PG-SGA score ≥9. 7. Inability to comprehend trial requirements or likelihood of non-compliance with trial requirements.

  8. Presence of hematogenous metastases. 9. Presence of other malignant lesions, excluding curable non-melanoma skin cancer, cervical carcinoma in situ, or malignancies with a cure ≥5 years.

  10. Known grade 3 to 4 allergic reactions to any treatment component. 11. Participation in other clinical trials within the past 30 days. 12. Active autoimmune diseases or history of autoimmune diseases (such as interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism); exceptions include vitiligo or resolved atopic asthma without the need for intervention in adulthood; patients with stable doses of thyroid replacement hormone therapy for autoimmune-mediated hypothyroidism and patients with stable doses of insulin for type I diabetes can be included.

  13. History of immunodeficiency, including HIV-positive status, or other acquired or congenital immunodeficiency diseases, or history of organ transplantation and allogeneic bone marrow transplantation.

  14. Uncontrolled clinical symptoms or diseases of the heart, such as (1) NYHA class II or higher heart failure (2) Unstable angina (3) Myocardial infarction within the past year (4) Clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention.

  15. Active pulmonary tuberculosis infection detected by history or CT examination, or history of active pulmonary tuberculosis infection within the past year before enrollment, or history of active pulmonary tuberculosis infection more than 1 year ago without proper treatment.

  16. Presence of active hepatitis B (HBV DNA ≥ 2000 IU/mL or 1× 104 copies/mL), hepatitis C (positive HCV antibodies, and HCV-RNA higher than the detection limit of the assay).

  17. According to the investigator's judgment, concurrent diseases that pose a serious risk to patient safety or may interfere with patient completion of the study, or other reasons deemed unsuitable for enrollment by the investigator.

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 191 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
mPFS | The time from the start of treatment, for half of the participants in a study to experience disease progression or death from any cause
  Median Progression-free survival (PFS) assessed in the intention-to-treat (ITT) population according to RECIST 1.1 criteria.

SECONDARY OUTCOMES:
OS | occurence or end of follow-up（2 years after enrollment）, which comes first
  The length of time from the start of treatment until the point of death from any cause.
ORR | 2 months after enrollment
  objective response rate
DoR | occurence or end of follow-up（2 years after enrollment）, which comes first
  Duration of Response

CONTACTS AND LOCATIONS:
Overall Officials: Yongling Ji, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No